CLINICAL TRIAL: NCT04024150
Title: Impact of in Utero Exposure to Anti-integrase Antiretrovirals on the Newborn Immune System
Brief Title: Pregnancy, Anti-integrase and Lymphocyte Repertoire of the Newborn
Acronym: RAGIIF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190394; 2019-A00926-51 (Other: ID RCB number)
Record Dates: First submitted 2019-07-02; First posted 2019-07-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Anti-integrases
Keywords: Anti-integrases treatment; Antiretroviral treatment; Pregnancy
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Newborns exposed: Newborns exposed in-utero to raltegravir
  Interventions: Biological: Blood test
- Newborns controls: Newborns exposed to antiretroviral therapy without anti-integrase
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — Single blood sample of 2 ml at birth on the occasion of blood sampling routine checkup

SUMMARY:
The objective of the study is to evaluate at birth, the diversity of the T repertoire of newborns exposed in utero to anti-integrases in comparison with a control group of children exposed to other antiretroviral drugs.

DETAILED DESCRIPTION:
Antiretroviral treatment during pregnancy is remarkably effective in preventing the transmission of mother-to-child viruses. Molecules of the class of anti-integrases are still little used during pregnancy, but their prescription is increasing given their intrinsic effectiveness and their overall tolerance profile.

The integrase of HIV-1, responsible for the integration of viral DNA in cellular DNA, has a functional similarity with human RAG1 / 2 proteins, responsible for V (D) J recombination. RAG1 / 2 proteins alteration is associated in human clinic with immune disturbances of varied severity.

The objective of the study is to evaluate at birth, the diversity of the T repertoire of newborns exposed in utero to anti-integrases in comparison with a control group of children exposed to other antiretroviral drugs.

ELIGIBILITY:
Inclusion Criteria:

* No parental opposition after information. "Exposed" group :
* Newborn at term exposed to raltegravir (RTG) before 8 weeks of gestation and until the end of pregnancy. Children exposed to elvitegravir (ETG), dolutegravir (DTG) or bictegravir (BTG) may be included but will be analyzed separately.

"Control" group :

- Term neonate exposed to antiretroviral therapy without anti-integrase.

Exclusion Criteria:

* Prematurity less than 36 weeks of gestation.
* Organ dysfunction.
* Acute or chronic fetal distress, need for hospitalization in neonatology, malformation syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborns exposed in utero to an antiretroviral therapy and born in the maternities of Paris AP-HP hospitals: Necker, Pitié-Salpétrière, Bichat, Louis Mourier and Cochin (Port-Royal).
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Newborn immunity | 18 months
  T cells immune repertoire integrity

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Blanche, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Jean-Pierre de Villartay, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (5):
- France (5):
  - AP-HP, Hôpital Louis Mourier, Colombes
  - AP-HP, Hôpital de la Pitié Salpêtrière, Paris
  - AP-HP, Hôpital Cochin, Paris
  - AP-HP, Hôpital Necker, Paris
  - AP-HP, Hôpital Bichat-Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Villartay JP, Pannier E, Sibiude J, Frange P, Tubiana R, Blanche S. Brief Report: T-Cell Receptor alpha Repertoire Diversity at Birth After in utero Exposure to HIV Integrase Strand-Transfer Inhibitors. J Acquir Immune Defic Syndr. 2023 Mar 1;92(3):260-262. doi: 10.1097/QAI.0000000000003130. PMID 36343360